CLINICAL TRIAL: NCT00740324
Title: Exploratory Study of Additional Use of Scopolamine Butylbromide, Glucagon or NPO-11 Following Single Dose of NPO-11 in Healthy Adult Men During Endoscopy
Brief Title: Exploratory Study of Additional Use of Scopolamine Butylbromide, Glucagon or NPO-11 Following Single Dose of NPO-11 in Healthy Adult Men
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nihon Pharmaceutical Co., Ltd (Industry)
Responsible Party: Yasumasa Ogawa, Nihon Pharmaceutical Co., Ltd
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NPO-11-01/SE-02
Record Dates: First submitted 2008-08-21; First posted 2008-08-22 (Estimated); Last update posted 2010-11-09 (Estimated); Status verified 2010-11

CONDITIONS: Healthy
Keywords: During; Endoscopy; Gastric; Peristalsis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- N (Active Comparator)
  Interventions: Drug: NPO-11
- B (Active Comparator)
  Interventions: Drug: NPO-11
- G (Active Comparator)
  Interventions: Drug: NPO-11

INTERVENTIONS:
Drug: NPO-11 — 20 mg butylscopolammonium bromide after administration of NPO-11
  Arms: B
Drug: NPO-11 — NPO-11 after administration of NPO-11
  Arms: N
Drug: NPO-11 — 1 mg glucagons after administration of NPO-11
  Arms: G

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of the additional administration of scopolamine butylbromide, glucagon or NPO-11 following a single intragastric dose of NPO-11 during endoscopy in healthy adult men. The safety will be evaluated based on adverse events and adverse drug reactions (ADRs) observed with NPO-11 + scopolamine butylbromide or glucagon, and following additional administration of NPO-11. The efficacy will be evaluated based on changes in the frequency of gastric peristalsis classification after the initial dose and the additional dose, and on the presence or absence of gastric peristalsis at each evaluation point.

ELIGIBILITY:
Inclusion Criteria:

Healthy adult male volunteers who meet all the following criteria will be enrolled in the study. Subjects have to provide written informed consent for voluntary participation in the study.

1. Volunteers who are in good health as confirmed by the investigator or subinvestigator
2. Volunteers (age from 35 to less than 65 years old at the time of consent)

Exclusion Criteria:

Volunteers who meet any of the following criteria will be excluded from the study.

1. Volunteers with any clinically significant symptoms, physical findings or laboratory values at screening visit which are considered unsuitable for participation in the study in the investigator's or subinvestigator's opinion
2. Volunteers with a history of surgery in the upper gastrointestinal tract
3. Volunteers with a history of shock or hypersensitivity to l-menthol or peppermint oil (mint oil)
4. Volunteers with a history of shock or hypersensitivity to scopolamine butylbromide, glucagon, lidocaine hydrochloride or heparin sodium
5. Volunteers who are contraindicated for administration of scopolamine butylbromide or glucagon in the investigator's or subinvestigator's opinion based on health interview
6. Volunteers who have been exposed to NPO-11
7. Volunteers who have received other investigational drugs within four months before consent or who are participating in other clinical studies
8. Volunteers otherwise ineligible for participation in the study in the investigator's or subinvestigator's opinion

Ages: 35 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2008-08; Primary Completion 2009-03 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
[Safety] (Evaluation by investigator or subinvestigator) Adverse events and ADRs observed between administration and 7 ± 3 days after administration | 7 ± 3 days after administration

SECONDARY OUTCOMES:
[Efficacy] (Central evaluation by independent evaluator) (1) Change in the frequency of gastric peristalsis classification (2) Presence or absence of gastric peristalsis at each evaluation point | each evaluation point

CONTACTS AND LOCATIONS:
Locations (1):
- Tokyo, Japan